CLINICAL TRIAL: NCT05584696
Title: Effectiveness of Green Color Exposure on Dental Anxiety for Third Molar Surgery
Brief Title: Effectiveness of Green Color Exposure on Dental Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Gokhan Gurses, Assistant Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SelcukU001
Record Dates: First submitted 2022-09-27; First posted 2022-10-18 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Anxiety, Dental; Post Operative Pain
MeSH Terms: conditions — Anxiety Disorders; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Green Light Exposure Group (Experimental): When patients enter the clinic, toss a coin to determine which group they will belong to. Before the patient puts on the green glasses, the anxiety level is measured with the help of VAS. Then the patient is seated in the dental unit and green glasses will be put on. After 10 minutes the anxiety level will be measured again with the help of VAS.
  The level of pain felt during surgery was determined by VAS. All operations will be performed by a single experienced surgeon. Since the patients enter the clinic, their heart rate, oxygen saturation and blood pressure will be measured continuously.
  Interventions: Other: Green light exposure
- Control Group (Placebo Comparator): When patients enter the clinic, toss a coin to determine which group they will belong to. Before the patient puts on transparent glasses, the anxiety level is measured with the help of VAS. Then the patient is seated in the dental unit and transparent glasses will be put on. After 10 minutes the anxiety level will be measured again with the help of VAS.
  The level of pain felt during surgery was determined by VAS. All operations will be performed by a single experienced surgeon. Since the patients enter the clinic, their heart rate, oxygen saturation and blood pressure will be measured continuously.
  Interventions: Other: Normal light exposure

INTERVENTIONS:
Other: Green light exposure — The experimental group wears green color glasses ten minutes before surgery until it ends.
  Arms: Green Light Exposure Group
Other: Normal light exposure — The control group wears green color glasses ten minutes before surgery until it ends.
  Arms: Control Group

SUMMARY:
The investigator's aim in this study was to evaluate the preoperative anxiety and the pain felt during the operation due to exposure to green light. For this purpose, the participants will wear green or translucent glasses before the operation. The investigator will evaluate the patient's anxiety change and the pain she/he feels during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 and ASA 2 patient population
* not having had a third molar surgery before
* volunteer to participate in the study

Exclusion Criteria:

* dental phobia
* patients who will be treated under general anesthesia
* refusing the measurements
* not filling the VAS

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
Pre-op Anxiety Score-1(VAS) | 1 minute after the participant enters the clinic
  Patients fill out the Dental Anxiety Scale(Visual Analogue Scale) when he/she arrives dental clinic. The range of Scala is 0-10. A lower score means better results.
Pre-op Anxiety Score-1(STAI-State) | 1 minute after the participant enters the clinic
  Patients fill out the State-Trait Anxiety Inventory-State when he/she arrives dental clinic. The range of Scala is 0-10. A lower score means better results.
Pre-op Anxiety Score-2(VAS) | 10 minutes after the glasses put on
  Patients fill out the Dental Anxiety Scale(Visual Analogue Scale) ten minutes after wearing green or translucent glasses in the dental unit. The range of Scala is 0-10. A lower score means better results.
Pre-op Anxiety Score-2(STAI-State) | 10 minutes after the glasses put on
  Patients fill out the State-Trait Anxiety Inventory-State ten minutes after wearing green or translucent glasses in the dental unit. The range of Scala is 0-10. A lower score means better results.
Pre-op blood pressure-1 | 1 minute after the participant enters the clinic
  Brachial tension measurement. ideally it should be 120-80 mm/hg. Çeviri sonuçları After the patient enters the clinic
Pre-op blood pressure-2 | 10 minutes after the glasses are put on
  Brachial tension measurement. ideally it should be 120-80 mm/hg.
Pre-op blood oxygen level-1 | 1 minute after the participant enters the clinic
  saturation measurement from finger tip by pulse oximeter. The avarage value is above %90.
Pre-op blood oxygen level-2 | 10 minutes after the glasses are put on
  saturation measurement from finger tip by pulse oximeter. The avarage value is above %90.
Pre-op Pulsation-1 | 1 minute after the participant enters the clinic
  heartbeat measurement by pulse oximeter. The avarage value is between 65-75.
Pre-op Pulsation-2 | 10 minutes after the glasses are put on and the patient sits in the chair
  heartbeat measurement by pulse oximeter. The avarage value is between 65-75.
Intraoperative Pain Score | 1 minutes after
  Measuring the pain felt by the patient after the operation with the help of the visual analog scale. The range of Scala is 0-10. A lower score means better results.

CONTACTS AND LOCATIONS:
Overall Officials: Gökhan Gürses, Study Chair — Selcuk University, Faculty of Dentistry
Locations (1):
- Selcuk University, Faculty of Dentistry, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gurses G, Omeroglu Akkoc FI, Akti A, Korez MK. Effectiveness of wearing glasses with green lenses on dental anxiety for third-molar surgery: A randomized clinical trial. J Am Dent Assoc. 2024 Jun;155(6):496-503.e1. doi: 10.1016/j.adaj.2024.02.006. Epub 2024 Mar 21. PMID 38520420